CLINICAL TRIAL: NCT05445128
Title: A Phase 2, Open-Label Study to Evaluate the Efficacy and Safety of MGTA-145 in Combination With Plerixafor for the Mobilization of Hematopoietic Stem Cells in Patients With Sickle Cell Disease
Brief Title: Study of MGTA-145 and Plerixafor in Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was voluntarily terminated due to a business decision not to proceed, and not due to any safety issue.
Sponsor: Ensoma (Industry)
Collaborators: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 145-SCD-204
Record Dates: First submitted 2022-05-26; First posted 2022-07-06 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-01

CONDITIONS: Sickle Cell Disease
Keywords: SCD; MGTA-145; Plerixafor; Mobilization; Apheresis
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single Day Dosing/Apheresis (Experimental): Single dose of MGTA-145 in combination with plerixafor followed by apheresis
  Interventions: Biological: MGTA-145; Drug: Plerixafor
- Part B: 2-Day Dosing/Apheresis (Experimental): MGTA-145 in combination with plerixafor followed by apheresis on two consecutive days
  Interventions: Biological: MGTA-145; Drug: Plerixafor

INTERVENTIONS:
Biological: MGTA-145 — MGTA-145 will be administered as an IV infusion
Drug: Plerixafor — 240 µg/kg administered subcutaneously

SUMMARY:
This research study is designed to investigate a new potential medicine for mobilizing stem cells and apheresis collection in patients with Sickle Cell Disease. MGTA-145, the new potential medicine, will be given with plerixafor.

DETAILED DESCRIPTION:
This Phase 2, multicenter, open-label study will be conducted in 2 parts (Parts A and B). Part A is intended to characterize the efficacy, safety, PK and PD of a single dose of MGTA-145 and plerixafor for HSC mobilization and apheresis collection in patients with SCD. Part B is designed to characterize the efficacy, safety, PK and PD of 2 consecutive days of dosing with MGTA-145 and plerixafor for HSC mobilization and apheresis collection in patients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 to ≤35 years of age.
* Subject must weigh ≥30 kg.
* Subject must have a diagnosis of Sickle Cell Disease.

Exclusion Criteria:

* Subject must not have had a vaso-occlusive event (VOE) requiring a visit to a healthcare facility within 30 days of screening.
* Subject must not have undergone or attempted and failed previous hematopoietic stem cell (HSC) collection.
* Subject must not have had a prior autologous or allogeneic transplantation, inclusive of gene therapy.
* Male subject must be willing or able to use a highly effective method of contraception for 3 months during and after treatment.
* Female subject must not be pregnant or breastfeeding. If sexually active, female subject must be willing or able to use a highly effective method of contraception for 3 months during and after treatment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hyun Lee, MD, MPH, Study Director — Magenta Therapeutics
Locations (3):
- United States (3):
  - National Institutes of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated early by original sponsor after first patient dosed. Only 1 participant was enrolled in Part A and no participants were enrolled in Part B.
Period: Overall Study
Arm/Group | Part A: Single Day Dosing/Apheresis | Part B: 2-Day Dosing/Apheresis
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apheresis Collection Yield
Description: Determination of the yield of CD34+ cells after either one or two consecutive days of MGTA-145 and plerixafor mobilization followed by apheresis.
Time Frame: Up to 2 days
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 0

2. Primary Outcome: Assess Number of Participants With Treatment Emergent Adverse Events Leading to Study Drug Discontinuation Based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Description: Assess number of participants with treatment emergent adverse events leading to study drug discontinuation based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 30 days
Population: Study terminated early by original sponsor after first patient dosed
Measure: Number; unit: participants
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 1
participants | 0

3. Primary Outcome: Assess the Number of Participants With Treatment Emergent >/= Grade 3 Clinical Laboratory Abnormalities Based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Description: Assess the number of participants with treatment emergent >/= Grade 3 clinical laboratory abnormalities based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 11 days
Population: Study terminated early by original sponsor after first patient dosed
Measure: Number; unit: participants
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 1
participants | 0

4. Primary Outcome: Vital Signs - Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital Signs - Number of participants with clinically significant changes from baseline in vital signs
Time Frame: Up to 11 days
Population: Study terminated early by original sponsor after first patient dosed
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Laboratory Assessment - Number of Participants With Clinically Significant Changes From Baseline in Hematology and Clinical Chemistry Laboratory Parameters.
Description: Laboratory Assessment - Number of participants with clinically significant changes from baseline in hematology and clinical chemistry laboratory parameters.
Time Frame: Up to 11 days
Population: Study terminated early by original sponsor after first patient dosed
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 1
Participants | 1

6. Secondary Outcome: Mobilization Effects of Single-day and Two-day Dosing With MGTA-145 and Plerixafor in Peripheral Blood in Patients With SCD
Description: Determination of peak peripheral blood CD34+ counts single-day and two-day dosing with MGTA-145 and plerixafor in peripheral blood in patients with SCD
Time Frame: Up to 2 days
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 0

7. Secondary Outcome: Investigate Plasma Concentrations of MGTA-145 Per Timepoint of Collection (Pharmacokinetics)
Description: Investigate plasma concentrations of MGTA-145 per timepoint of collection (Pharmacokinetics)
Time Frame: Up to 2 days
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 0

8. Secondary Outcome: Assess Presence of MGTA-145 Anti-Drug Antibodies (ADA) in Plasma Samples (Using Electrochemiluminescent Immunoassay [ECLIA])
Description: Assess presence of MGTA-145 Anti-Drug Antibodies (ADA) in plasma samples (using electrochemiluminescent immunoassay [ECLIA])
Time Frame: Up to 11 days
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 0

9. Secondary Outcome: Assess Titers of MGTA-145 Anti-Drug Antibodies (ADA) in Plasma Samples (Using Electrochemiluminescent Immunoassay [ECLIA])
Description: Assess titers of MGTA-145 Anti-Drug Antibodies (ADA) in plasma samples (using electrochemiluminescent immunoassay [ECLIA])
Time Frame: Up to 11 days
Population: Study terminated early by original sponsor after first patient dosed
Arm/Group | Part A: Single Day Dosing/Apheresis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Arm/Group | Part A: Single Day Dosing/Apheresis
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Single Day Dosing/Apheresis (N=1)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Study terminated early by original sponsor after first patient dosed. Only 1 participant was enrolled in Part A and no participants were enrolled in Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT05445128/Prot_000.pdf